CLINICAL TRIAL: NCT04605159
Title: A Phase III, Randomized, Double-blind, Placebo-controlled Multi-country Study to Demonstrate Efficacy of a Single Dose of Unadjuvanted RSV Maternal Vaccine, Administered IM to Pregnant Women 18 to 49 Years of Age, for Prevention of RSV Associated LRTIs in Their Infants up to 6 Months of Age
Brief Title: A Phase III, Double-blind Study to Assess Safety and Efficacy of an RSV Maternal Unadjuvanted Vaccine, in Pregnant Women and Infants Born to Vaccinated Mothers
Acronym: GRACE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Following a recommendation from the Independent Data Monitoring Committee of NCT04605159 (RSV MAT 009), GSK made the decision to stop enrolment and vaccination in the study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 212171; 2020-001355-40 (EudraCT Number)
Record Dates: First submitted 2020-10-22; First posted 2020-10-27 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Following the decision to stop enrollment and vaccination, the study/site staff and maternal participants no longer stayed blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- RSV MAT Group - Mother (Experimental): Maternal participants received a single dose of the RSV MAT vaccine administered at Day 1 in this study.
  Interventions: Biological: RSV MAT
- Placebo Group - Mother (Placebo Comparator): Maternal participants received a single dose of placebo administered at Day 1 in this study.
  Interventions: Drug: Placebo
- RSV MAT Group - Infant (No Intervention): This group consisted of infants born to mothers (from RSV MAT Group - Mother) who received a single dose of RSV MAT vaccine during pregnancy.
- Placebo Group - Infant (No Intervention): This group consisted of infants born to mothers (from Placebo Group - Mother) who received a single dose of placebo during pregnancy.

INTERVENTIONS:
Biological: RSV MAT — One dose of RSV MAT vaccine reconstituted with NaCl solution, administered intramuscularly in the non-dominant arm at Day 1.
  Arms: RSV MAT Group - Mother
Drug: Placebo — One dose of placebo (lyophilized sucrose reconstituted with NaCl solution) administered intramuscularly in the non-dominant arm at Day 1.
  Arms: Placebo Group - Mother

SUMMARY:
The purpose of this study was to evaluate the ability of a single dose of the investigational RSV Maternal vaccine, administered intramuscularly (IM) to pregnant women aged 18-49 years, in good general maternal health, in preventing medically assessed RSV associated Lower Respiratory Tract Illnesses (LRTIs) in infants born to vaccinated mothers. The study also evaluated the safety of the investigational RSV Maternal vaccine both in vaccinated mothers and in their corresponding infant.

Following a recommendation from the Independent Data Monitoring Committee of NCT04605159 (RSV MAT 009), GSK made the decision to stop enrolment and vaccination in the study. Ongoing study participants at that time continued to be monitored as part of the study.

ELIGIBILITY:
Inclusion Criteria:

Maternal participants

* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Participants who give written or witnessed/thumb printed informed consent after the study has been explained, and before any study specific procedures are performed, as per local regulations regulatory requirements.
* Age 18 to 49 years, inclusive, at the time of study intervention.
* Pre-pregnancy BMI 17.0 to 39.9 kg/m2, inclusive.
* In good general maternal health as established by medical history and clinical examination before entering into the study.
* Singleton pregnancy (including instances where the singleton pregnancy derives from a vanishing twin syndrome).
* At 24^0/7 to 34^0/7 weeks of gestation at the time of study vaccination (Visit 1), as established by:
* last menstrual period (LMP) date corroborated by first or second trimester ultrasound examination (U/S) i.e. at or before 28 weeks of gestation.
* 1st or 2nd trimester U/S only, if LMP is unknown/uncertain
* Certain LMP, corroborated by an U/S performed after 28 weeks of gestation is also acceptable.
* No fetal genetic abnormalities (based on genetic testing, if performed).
* No significant congenital malformations, as assessed by fetal anomaly ultrasound scan conducted at or beyond 18 weeks of gestation.
* Willing to provide cord blood.
* Who do not plan to give their child for adoption.
* Who plan to reside in the study area for at least one year after delivery.
* Willing to have the infant followed-up after delivery for a period of 12 months.

Infant participants

* Live-born from the study pregnancy.
* If required per local regulations/guidelines, re-signed (confirmed) written or witnessed/thumb printed informed consent for study participation of the infant obtained from the infant's mother and/or father and/or LAR, before performing any study specific procedure. OR, if permitted by local regulation, documented verbal consent for infant's participation obtained from the parent(s)/LAR(s) at birth, followed by written consent obtained by (or before) Visit 2-newborn.

Exclusion Criteria:

Maternal participants Medical conditions

* History of allergic disease or reactions likely to be exacerbated by any component of the RSV vaccine
* Hypersensitivity to latex
* Significant complications in the current pregnancy:
* Gestational hypertension unless blood pressure it is controlled and maintained in the normal range (<140mmHg and <90mmHg) through diet and/or antihypertensive medications
* Gestational diabetes not controlled by medication, diet and/or exercise
* Pre-eclampsia
* Eclampsia
* Intrauterine Growth Restriction/Fetal Growth Restriction
* Placenta previa
* Placental abruption, placenta accreta/percreta/increta, chorioamnionitis or any abnormalities that can impair the maternal-fetal circulation
* Polyhydramnios
* Oligohydramnios
* Preterm labour or history of preterm labour in the current pregnancy
* Any intervention to prevent preterm delivery or medical treatment for suspected preterm delivery, including administration of systemic corticosteroids for fetal lung maturation
* Cholestasis
* Other pregnancy-related complications (per investigator's judgement)
* Significant structural abnormalities of the uterus or cervix
* History of 2 or more prior stillbirths or neonatal deaths/history of 2 or more preterm births at ≤34 weeks gestation/3 or more consecutive spontaneous abortions
* Known HIV infection (as per serological tests performed during the current pregnancy)
* Known or suspected HBV or HCV infection
* Known or suspected infection during the current pregnancy with Toxoplasma, Parvovirus B19, Syphilis, Zika, Rubella, Varicella, CMV or primary genital Herpes Simplex
* Active infection with tuberculosis
* Known or suspected impairment of the immune system
* Current autoimmune disorder for which the participant has received immune-modifying therapy within 6 months before study vaccination, or plans administration through delivery
* Lymphoproliferative disorder or malignancy within 5 years before study vaccination
* Acute or chronic clinically significant abnormality or poorly controlled pre-existent co-morbidities or any other clinical conditions that might pose additional risk to the participant due to participation in the study
* Any conditions that may interfere with participant's ability to comply with study procedures or receipt of prenatal care
* Any condition which would increase the risks of study participation to the unborn infant

Prior/Concomitant therapy

* Prior receipt of an RSV vaccine in the current pregnancy
* Use of any investigational/non-registered product other than the study vaccine/product as described below, or planned use during the period :
* For a drug, vaccine or medical device: from 29 days before the dose of study vaccine
* For immunoglobulins: 3 months before the dose of study vaccine/product.

The exception to this is investigational products administered in the setting of a pandemic which may be allowed following delivery

* Planned administration/administration of any vaccine from 29 days before the dose of study vaccine or planned administration through delivery, except:
* Seasonal influenza vaccines, tetanus vaccines, dTpa/Tdap - alone vaccines, dTpa/Tdap vaccines that also contain other antigens, Hepatitis B vaccines, and COVID-19 vaccines all of which may be administered according to standard of care ≥15 days before or after study vaccination
* Administration of immunoglobulins (except anti-Rh0D IG, which may be administered at any time), blood products or plasma derivatives within 3 months before study vaccination or planned administration through delivery
* Administration of immune-modifying therapy within 6 months before the study vaccination, or planned administration through delivery. This includes but is not limited to:
* Azathioprine, mycophenolate mofetil, 6-mercaptopurine, cyclosporine, tacrolimus, monoclonal or polyclonal antibodies
* Prednisone ≥5 mg/day or equivalent for ≥14 days; Inhaled, intra-articular/intra-bursal and topical steroids are allowed
* Corticosteroids administered for fetal lung maturation

Prior/Concurrent clinical study experience

- Concurrently participating in another clinical study, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product

Other exclusions

* Alcoholism or substance use disorder within the past 24 months based on DSM-5 criteria
* A local condition that precludes injection of the study vaccine/product or precludes assessment of local reactogenicity
* Consanguinity of maternal participant and her partner (second degree cousins or closer)
* Any study personnel or their immediate dependants, family or household members

Infant participants

* Concurrently participating in another clinical study, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product
* Any condition which would increase the risks of study participation to the infant
* Child in care.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11194 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (134):
- United States (38):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Blackfoot, Idaho
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Saginaw, Michigan
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Grand Island, Nebraska
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Englewood, Ohio
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Hendersonville, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Burleson, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Keller, Texas
  - GSK Investigational Site, Lampasas, Texas
  - GSK Investigational Site, League City, Texas
  - GSK Investigational Site, McAllen, Texas
  - GSK Investigational Site, Mesquite, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Weatherford, Texas
  - GSK Investigational Site, Norfolk, Virginia
- Argentina (4):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad AutOnoma de Buenos Aire
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (5):
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Southport, Queensland
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Bangladesh (2):
  - GSK Investigational Site, Matlab
  - GSK Investigational Site, Sylhet
- Belgium (5):
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Sint-Niklaas
- Brazil (6):
  - GSK Investigational Site, Caxias do Sul
  - GSK Investigational Site, Nova Iguaçu
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, RibeirAo PretoSP
  - GSK Investigational Site, Santa Maria
  - GSK Investigational Site, São José do Rio Preto
- Canada (4):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- Colombia (5):
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Cali Colombia
  - GSK Investigational Site, Chía
  - GSK Investigational Site, Medellín
- GSK Investigational Site, Santo Domingo Este, Dominican Republic
- Finland (5):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (5):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pierre-Bénite
- Honduras (2):
  - GSK Investigational Site, Comayagua
  - GSK Investigational Site, San Pedro Sula
- India (6):
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Mangalore
  - GSK Investigational Site, Mysore
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Vadu Budruk Pune
- Italy (7):
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Messina
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Novara
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Prato
  - GSK Investigational Site, Verona
- Mexico (6):
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Monterrey
  - GSK Investigational Site, Morelia
  - GSK Investigational Site, Oaxaca City
  - GSK Investigational Site, San Juan del Río
  - GSK Investigational Site, San Luis Potosí City
- New Zealand (3):
  - GSK Investigational Site, Grafton Auckland
  - GSK Investigational Site, Papatoetoe Auckland
  - GSK Investigational Site, Wellington
- GSK Investigational Site, Panama City, Panama
- Philippines (2):
  - GSK Investigational Site, Cavite
  - GSK Investigational Site, Manila
- South Africa (4):
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Soshanguve
  - GSK Investigational Site, Soweto
- South Korea (2):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Seoul
- Spain (13):
  - GSK Investigational Site, Aravaca
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Boadilla Del Monte Madrid
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Getafe
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Seville
  - GSK Investigational Site, TorrejOn Ardoz Madrid
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
- Taiwan (5):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- GSK Investigational Site, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Dieussaert I, Hyung Kim J, Luik S, Seidl C, Pu W, Stegmann JU, Swamy GK, Webster P, Dormitzer PR. RSV Prefusion F Protein-Based Maternal Vaccine - Preterm Birth and Other Outcomes. N Engl J Med. 2024 Mar 14;390(11):1009-1021. doi: 10.1056/NEJMoa2305478. PMID 38477988
- [Derived] Banooni P, Gonik B, Epalza C, Reyes O, Madhi SA, Gomez-Go GD, Zaman K, Llapur CJ, Lopez-Medina E, Stanley T, Kantele A, Huang LM, Mussi-Pinhata MM, Dewulf J, Langley JM, Seidl C, Ota M, Kirabo M, Anspach B, Dieussaert I, Henry O, Kim JH, Picciolato M. Efficacy, Immunogenicity, and Safety of an Investigational Maternal Respiratory Syncytial Virus Prefusion F Protein-Based Vaccine. Clin Infect Dis. 2026 Feb 9;82(1):e146-e155. doi: 10.1093/cid/ciaf033. PMID 39879629
- [Derived] Ginsburg AS, Srikantiah P. Respiratory syncytial virus: promising progress against a leading cause of pneumonia. Lancet Glob Health. 2021 Dec;9(12):e1644-e1645. doi: 10.1016/S2214-109X(21)00455-1. Epub 2021 Nov 11. No abstract available. PMID 34774184

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 11194 participants (5959 maternal participants and 5235 infants) completed the informed consent process, of which 5328 maternal participants were exposed to the study intervention, and 5235 infants were born to those exposed mothers (RSV MAT Group - Mother and Placebo Group - Mother). Therefore, 10563 participants started the study.
Period: Overall Study
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother | RSV MAT Group - Infant | Placebo Group - Infant
Started | 3557 | 1771 | 3494 | 1741
Completed | 3374 | 1657 | 3236 | 1583
Not Completed | 183 | 114 | 258 | 158
Not completed — Adverse Event | 6 | 3 | 21 | 4
Not completed — Lost to Follow-up | 74 | 45 | 119 | 80
Not completed — Protocol Violation | 4 | 5 | 2 | 0
Not completed — Withdrawal by Subject | 66 | 37 | 68 | 50
Not completed — Migrated / moved from the study area | 32 | 22 | 41 | 21
Not completed — Other | 1 | 2 | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother | RSV MAT Group - Infant | Placebo Group - Infant | Total
Number analyzed (Participants) | 3557 | 1771 | 3494 | 1741 | 10563
Age, Customized [Count of Participants; unit: Participants]
  0 to 1 years of age | 0 | 0 | 3494 | 1741 | 5235
  18 to 34 years of age | 2866 | 1408 | 0 | 0 | 4274
  35 to 39 years of age | 581 | 300 | 0 | 0 | 881
  40 to 49 years of age | 110 | 63 | 0 | 0 | 173
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 3557 | 1771 | 1739 | 867 | 7934
  Male | 0 | 0 | 1753 | 873 | 2626
  Other, Unspecified | 0 | 0 | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 663 | 326 | 641 | 321 | 1951
  BLACK OR AFRICAN AMERICAN | 517 | 251 | 463 | 234 | 1465
  WHITE | 1669 | 838 | 1634 | 816 | 4957
  OTHER, UNSPECIFIED | 685 | 345 | 730 | 348 | 2108
  OTHER, DEIDENTIFIED | 23 | 11 | 26 | 22 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Infant Participants With Medically Assessed, RSV-associated Lower Respiratory Tract Illnesses (LRTIs) of Any Severity and RSV-associated Severe LRTIs From Birth to Day 181 Post-birth
Description: An RSV-associated LRTI of any severity was characterized by a history of cough OR difficulty in breathing, AND a blood oxygen saturation by pulse oximetry (SpO2) lower than (<) 95%, OR respiratory rate increase AND a confirmed RSV infection. An RSV-associated severe LRTI met the case definition of RSV-LRTI AND was additionally characterized by a SpO2 <93%, OR lower chest wall in-drawing, OR inability to feed, OR failure to respond/unconscious. Medically assessed = the infant was evaluated by a healthcare professional for the LRTI.
Time Frame: From birth to Day 181 post-birth
Population: The analysis was performed on the Modified Full Analysis - Efficacy set for infants, which included all infant participants in the Exposed set who were born after at least 4 weeks of their maternal participants vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3426 | 1711
Participants
  RSV-associated LRTIs of any severity | 16 | 24
  RSV-associated severe LRTIs | 8 | 14

2. Primary Outcome: Number of Infant Participants With at Least One Serious Adverse Event (SAE) From Birth to Day 181 Post-birth
Description: An SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect or resulted in other situations that were considered serious per medical or scientific judgment. At least one SAE = occurrence of at least one SAE regardless of intensity grade or relation to vaccination.
Time Frame: From birth to Day 181 post-birth
Population: The analysis was performed on the Exposed Set for infants, which included the infants live-born to exposed maternal participants, whose parents/legally acceptable representative(s) (LARs) completed the informed consent process and signed the informed consent form.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3494 | 1741
Participants | 640 | 323

3. Primary Outcome: Number of Infant Participants With at Least One Adverse Event (AE) Leading to Study Withdrawal From Birth to Day 181 Post-birth
Description: A participant was considered a 'withdrawal' from the study when no study procedure has occurred, no follow-up has been performed and no further information has been collected for this participant from the date of withdrawal/last contact. Participants who were withdrawn from the study because of AEs were clearly distinguished from participants who were withdrawn for other reasons. Investigators followed participants who were withdrawn from the study as a result of an AE until the event was resolved. At least one AE leading to study withdrawal = occurrence of at least one AE leading to study withdrawal regardless of intensity grade or relation to vaccination.
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3494 | 1741
Participants | 19 | 4

4. Primary Outcome: Number of Infant Participants With at Least One Medically Attended AE (MAE) From Birth to Day 181 Post-birth
Description: An MAE is defined as an unsolicited AE, such as a symptom or illness, which required hospitalization, or emergency room visit, or visit to/by a health care provider. At least one MAE = occurrence of at least one MAE regardless of intensity grade or relation to vaccination.
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3494 | 1741
Participants | 2321 | 1135

5. Primary Outcome: Number of Infant Participants With at Least One SAE From Birth to Day 366 Post-birth
Description: as for outcome 2
Time Frame: From birth to Day 366 post-birth
Population: The analysis was performed on the Exposed Set for infants, which included the infants live-born to exposed maternal participants, whose parents/LARs completed the informed consent process and signed the informed consent form.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3494 | 1741
Participants | 731 | 371

6. Primary Outcome: Number of Infant Participants With at Least One AE Leading to Study Withdrawal From Birth to Day 366 Post-birth
Description: as for outcome 3
Time Frame: From birth to Day 366 post-birth
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3494 | 1741
Participants | 21 | 4

7. Primary Outcome: Number of Infant Participants With at Least One MAE From Birth to Day 366 Post-birth
Description: as for outcome 4
Time Frame: From birth to Day 366 post-birth
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3494 | 1741
Participants | 2706 | 1330

8. Secondary Outcome: Number of Infant Participants With RSV-associated Hospitalizations From Birth to Day 181 Post-birth
Description: RSV-associated hospitalization is defined as a confirmed RSV infection and hospitalized for acute medical condition. Hospitalization is defined as admission for observation or treatment based on the judgment of a health care provider.
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3426 | 1711
Participants | 14 | 14

9. Secondary Outcome: Number of Infant Participants With All-cause LRTIs From Birth to Day 181 Post-birth
Description: All-cause LRTI was characterized by history of cough OR difficulty in breathing, AND SpO2 < 95%, OR respiratory rate increase.
Time Frame: From birth to Day 181 post-birth
Population: The analysis was performed on the Modified Full Analysis - Efficacy set for infants, which included all the infant participants in the Exposed Set who were born after at least 4 weeks of their maternal participants vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3426 | 1711
Participants | 162 | 103

10. Secondary Outcome: Number of Infant Participants With All-cause LRTIs With Hospitalization From Birth to Day 181 Post-birth
Description: All-cause LRTI was characterized by history of cough OR difficulty in breathing, AND SpO2 < 95%, OR respiratory rate increase. Hospitalization is defined as admission for observation or treatment based on the judgment of a health care provider.
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3426 | 1711
Participants | 30 | 22

11. Secondary Outcome: Number of Infant Participants With Medically Assessed, RSV-associated Severe LRTIs From Birth to Day 366 Post-birth
Description: An RSV-associated LRTI of any severity was characterized by a history of cough OR difficulty in breathing, AND an SpO2 <95%, OR respiratory rate increase AND a confirmed RSV infection. An RSV-associated severe LRTI met the case definition of RSV-LRTI AND was additionally characterized by an SpO2 <93%, OR lower chest wall in-drawing, OR inability to feed, OR failure to respond/unconscious. Medically assessed = the infant was evaluated by a healthcare professional for the LRTI.
Time Frame: From birth to Day 366 post-birth
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3426 | 1711
Participants | 38 | 22

12. Secondary Outcome: Number of Infant Participants With Medically Assessed, RSV-associated LRTIs of Any Severity From Birth to Day 366 Post-birth
Description: An RSV-associated LRTI of any severity was characterized by a history of cough OR difficulty in breathing, AND an SpO2 <95%, OR respiratory rate increase AND a confirmed RSV infection. Medically assessed = the infant was evaluated by a healthcare professional for the LRTI.
Time Frame: From birth to Day 366 post-birth
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3426 | 1711
Participants | 67 | 43

13. Secondary Outcome: Number of Infant Participants With Medically Assessed, RSV-associated Severe LRTIs for RSV Subtype A and RSV Subtype B Separately From Birth to Day 181 Post-birth
Description: An RSV-associated LRTI of any severity was characterized by a history of cough OR difficulty in breathing, AND an SpO2 <95%, OR respiratory rate increase AND a confirmed RSV infection. An RSV-associated severe LRTI met the case definition of RSV-LRTI AND was additionally characterized by an SpO2 <93%, OR lower chest wall in-drawing, OR inability to feed, OR failure to respond/unconscious. Medically assessed = the infant was evaluated by a healthcare professional for the LRTI. The RSV subtypes assessed for this analysis were RSV subtype A and RSV subtype B.
Time Frame: From birth to Day 181 post-birth
Population: The analysis was performed on the Modified Full Analysis - Efficacy set for infants which included all the infant participants in the Exposed Set who were born after at least 4 weeks of their maternal participants vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3426 | 1711
Participants
  RSV A | 2 | 3
  RSV B | 6 | 11

14. Secondary Outcome: Number of Infant Participants With Medically Assessed, RSV-associated LRTIs of Any Severity for RSV Subtype A and RSV Subtype B Separately From Birth to Day 181 Post-birth
Description: An RSV-associated LRTI of any severity was characterized by a history of cough OR difficulty in breathing, AND an SpO2 <95%, OR respiratory rate increase AND a confirmed RSV infection. Medically assessed = the infant was evaluated by a healthcare professional for the LRTI. The RSV subtypes assessed for this analysis were RSV subtype A and RSV subtype B.
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3426 | 1711
Participants
  RSV A | 6 | 8
  RSV B | 10 | 16

15. Secondary Outcome: Number of Infant Participants With Medically Assessed, RSV-associated Severe LRTIs From Birth to Day 121 Post-birth
Description: as for outcome 11
Time Frame: From birth to Day 121 post-birth
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3426 | 1711
Participants | 6 | 9

16. Secondary Outcome: Number of Infant Participants With Medically Assessed, RSV-associated LRTIs of Any Severity From Birth to Day 121 Post-birth
Description: as for outcome 12
Time Frame: From birth to Day 121 post-birth
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3426 | 1711
Participants | 9 | 15

17. Secondary Outcome: Number of Infant Participants With All-cause Pneumonia From Birth to Day 181 Post-birth
Description: The number of infant participants with all-cause pneumonia is presented in this outcome measure.
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3426 | 1711
Participants | 36 | 17

18. Secondary Outcome: Number of Infant Participants With RSV-associated Hospitalizations From Birth to Day 366 Post-birth
Description: as for outcome 8
Time Frame: From birth to Day 366 post-birth
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3426 | 1711
Participants | 41 | 26

19. Secondary Outcome: Number of Maternal Participants With RSV-associated Medically Attended RTIs (RSV-MA-RTIs) From Study Intervention Administration (Day 1) to Day 181 Post-delivery
Description: RSV-associated MA-RTI is defined as a medically attended visit for RTI symptoms and confirmed RSV infection.
Time Frame: From study intervention administration (Day 1) to Day 181 post-delivery
Population: The analysis was performed on the Exposed Set for maternal participants, which included all maternal participants who received the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother
Number analyzed (Participants) | 3557 | 1771
Participants | 3 | 6

20. Secondary Outcome: RSV-A Neutralizing Antibody Titers for Maternal Participants at Day 1, at Day 31 and at Delivery
Description: RSV-A neutralizing titers were determined by neutralization assay and expressed as geometric mean titers (GMTs).
Time Frame: At Day 1 (before study intervention administration), at Day 31 and at delivery
Population: The analysis was performed on the Per Protocol - Immunogenicity set for maternal participants, which included all maternal participants who received the study intervention to which they were randomized and had post-vaccination immunogenicity data available for the specified analysis at each of the specified time points (i.e. Day 1, Day 31, delivery) minus those participants with protocol deviations that led to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother
Number analyzed (Participants) | 404 | 196
Titers
  Day 1 | 637.2 [589.4 to 688.8] | 594.9 [527.3 to 671.2]
  Day 31: number analyzed (Participants) | 317 | 148
  Day 31 | 9196.9 [8310.8 to 10177.6] | 673.5 [578.8 to 783.7]
  Delivery: number analyzed (Participants) | 404 | 178
  Delivery | 5703.1 [5196.3 to 6259.3] | 657.7 [575.4 to 751.8]

21. Secondary Outcome: RSV-A Neutralizing Antibody Titers for Infant Participants at Delivery or Within 72 Hours After Birth
Description: RSV-A neutralizing titers were determined by neutralization assay and expressed as GMTs. The titers were measured on the cord blood sample collected at delivery, or on a blood sample collected from the infant within 72 hours after birth (if no cord blood sample could be obtained).
Time Frame: At delivery or within 72 hours after birth
Population: The analysis was performed on the Per Protocol - Immunogenicity set for infants, which included all infant participants in the Exposed set who had post-delivery/birth immunogenicity data available for the specified analysis at the specified time points (i.e. at delivery or within 72 hours after birth), minus those who (a) were born less than 4 weeks post- maternal participant vaccination and/ or (b) had protocol deviations that led to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 197 | 82
Titers | 9466.2 [8398.6 to 10669.5] | 725.9 [593.1 to 888.5]

22. Secondary Outcome: RSV-A Neutralizing Antibody Titers for Infant Participants at Day 43 Post-birth
Description: RSV-A neutralizing titers were determined by neutralization assay and expressed as GMTs.
Time Frame: At Day 43 post-birth
Population: The analysis was performed on a sub-cohort from the Per Protocol - Immunogenicity set for infants, which included the infant participants for whom blood samples were collected for the specified analysis at Day 43 post-birth.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 140 | 67
Titers | 4042.1 [3530.3 to 4628.2] | 311.3 [250.3 to 387.2]

23. Secondary Outcome: RSV-A Neutralizing Antibody Titers for Infant Participants at Day 121 Post-birth
Description: RSV-A neutralizing titers were determined by neutralization assay and expressed as GMTs.
Time Frame: At Day 121 post-birth
Population: The analysis was performed on a sub-cohort from the Per Protocol - Immunogenicity set for infants, which included the infant participants for whom blood samples were collected for the specified analysis at Day 121 post-birth.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 50 | 23
Titers | 682.4 [520.2 to 895.3] | 74.8 [46.5 to 120.2]

24. Secondary Outcome: RSV-A Neutralizing Antibody Titers for Infant Participants at Day 181 Post-birth
Description: RSV-A neutralizing titers were determined by neutralization assay and expressed as GMTs.
Time Frame: At Day 181 post-birth
Population: The analysis was performed on a sub-cohort from the Per Protocol - Immunogenicity set for infants, which included the infant participants for whom blood samples were collected for the specified analysis at Day 181 post-birth.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 44 | 9
Titers | 506.0 [432.4 to 592.3] | 133.7 [52.4 to 341.2]

25. Secondary Outcome: RSV MAT Immunoglobulin G (IgG)-Specific Antibody Concentrations for Maternal Participants at Delivery
Description: RSV MAT IgG-specific antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs) in ELISA units per milliliter (ELU/mL).
Time Frame: At delivery
Population: The analysis was performed on the Per Protocol - Immunogenicity set for maternal participants, which included all maternal participants who received the study intervention to which they were randomized and had post-vaccination immunogenicity data available for the specified analysis at the specified time point (i.e. delivery) minus those participants with protocol deviations that led to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother
Number analyzed (Participants) | 405 | 178
ELU/mL | 62880 [58517 to 67568] | 5600 [4949 to 6338]

26. Secondary Outcome: RSV MAT IgG-specific Antibody Concentrations for Infant Participants at Delivery or Within 72 Hours After Birth
Description: RSV MAT IgG-specific antibody concentrations were determined by ELISA and expressed as GMCs in ELU/mL. The antibody concentrations were measured on the cord blood sample collected at delivery, or on a blood sample collected from the infant within 72 hours after birth (only if no cord blood sample could be obtained at delivery).
Time Frame: At delivery or within 72 hours after birth (only if no cord blood sample could be obtained at delivery)
Population: The analysis was performed on the Per Protocol - Immunogenicity set for infants, which included all infant participants in the Exposed set who had post-delivery/birth immunogenicity data available for the specified analysis at the specified time points (i.e. at delivery or within 72 hours after birth), minus those who (a) were born less than 4 weeks post-maternal participant vaccination and/ or (b) had protocol deviations that led to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 230 | 97
ELU/mL | 94365 [86569 to 102864] | 6610 [5688 to 7682]

27. Secondary Outcome: Geometric Mean Ratio (GMR) Between Cord Blood and Maternal RSV MAT Immunoglobulin G (IgG)-Specific Antibody Concentrations
Description: The placental transfer ratio of RSV-MAT IgG-specific antibody concentration was determined from cord blood over that of the blood sample from mother at delivery. If no cord blood could be obtained, an infant blood sample was collected 72 hours after birth.
Time Frame: At delivery (for maternal participants) or within 72 hours after birth (for infant participants, only if no cord blood could be obtained)
Population: The analysis was performed on all pairs of maternal participants (from Per Protocol -Immunogenicity set for maternal participants) and their infants (from Per Protocol - Immunogenicity set for infants) with available results for this outcome measure at the specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- RSV MAT Group: This group consisted of pairs of maternal participants from RSV MAT Group - Mother and infant participants from RSV MAT Group - Infant.
- Placebo Group: This group consisted of pairs of maternal participants from Placebo Group - Mother and infant participants from Placebo Group - Infant.
Arm/Group | RSV MAT Group | Placebo Group
Number analyzed (Participants) | 150 | 60
Ratio | 1.46 [1.35 to 1.58] | 1.39 [1.22 to 1.59]

28. Secondary Outcome: Number of Maternal Participants With Any Solicited Administration Site Events From Day 1 to Day 7 Included
Description: Assessed solicited administration site events included erythema, pain and swelling at the injection site. Any pain = occurrence of the symptom regardless of intensity grade. Any erythema and swelling = symptom reported with a surface diameter greater than or equal to 20 millimeters.
Time Frame: From Day 1 to Day 7 included
Population: The analysis was performed on the Solicited Safety set for maternal participants, which included all maternal participants who received the study intervention and who had solicited safety data available during the specified period (i.e. from Day 1 to Day 7 included).
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother
Number analyzed (Participants) | 3090 | 1547
Participants
  Any Erythema | 133 | 8
  Any Pain | 1294 | 230
  Any Swelling | 96 | 8

29. Secondary Outcome: Number of Maternal Participants With Any Solicited Systemic Events From Day 1 to Day 7 Included
Description: Assessed solicited systemic events included abdominal pain, diarrhea, fatigue, headache, nausea, fever [temperature equal to or above (>=) 38 degrees Celsius (°C)/100.4 degrees Fahrenheit (°F), regardless of the location of measurement] and vomiting. Any = occurrence of the adverse event regardless of intensity grade or relation to study vaccination.
Time Frame: From Day 1 to Day 7 included
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother
Number analyzed (Participants) | 3090 | 1547
Participants
  Any Abdominal pain | 492 | 231
  Any Diarrhea | 351 | 180
  Any Fatigue | 1091 | 479
  Any Headache | 942 | 442
  Any Nausea | 599 | 306
  Any Fever | 26 | 7
  Any Vomiting | 276 | 149

30. Secondary Outcome: Number of Maternal Participants With Any Unsolicited AEs From Day 1 to Day 30 Included
Description: An unsolicited AE is defined as any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited AE. Any = occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: From Day 1 to Day 30 included
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother
Number analyzed (Participants) | 3557 | 1771
Participants | 629 | 297

31. Secondary Outcome: Number of Maternal Participants With at Least One SAE From Day 1 to Day 181 Post-delivery
Description: An SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant or resulted in abnormal pregnancy outcomes or in other situations that were considered serious per medical or scientific judgment. At least one SAE = occurrence of at least one SAE regardless of intensity grade or relation to vaccination.
Time Frame: From Day 1 to Day 181 post-delivery
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother
Number analyzed (Participants) | 3557 | 1771
Participants | 827 | 395

32. Secondary Outcome: Number of Maternal Participants With at Least One AE Leading to Study Withdrawal From Day 1 to Day 181 Post-delivery
Description: as for outcome 3
Time Frame: From Day 1 to Day 181 post-delivery
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother
Number analyzed (Participants) | 3557 | 1771
Participants | 6 | 3

33. Secondary Outcome: Number of Maternal Participants With at Least One All-cause MA-RTI From Day 1 to Day 181 Post-delivery
Description: All-cause MA-RTI occurred when the maternal participant visited a healthcare professional (e.g., a General Practitioner) for any respiratory symptom, including (but not limited to) cough, sore throat, sputum production and difficulty breathing. At least one all-cause MA-RTI = occurrence of at least one all-cause MA-RTI regardless of intensity grade or relation to vaccination.
Time Frame: From Day 1 to Day 181 post-delivery
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother
Number analyzed (Participants) | 3557 | 1771
Participants | 317 | 144

34. Secondary Outcome: Number of Maternal Participants With at Least One MAE From Day 1 to Day 42 Post-delivery
Description: as for outcome 4
Time Frame: From Day 1 to Day 42 post-delivery, an average of 2 months
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother
Number analyzed (Participants) | 3557 | 1771
Participants | 1717 | 785

35. Secondary Outcome: Number of Maternal Participants With Pregnancy Outcomes From Day 1 to Day 42 Post-delivery
Description: Assessed pregnancy outcomes included live birth with no congenital anomalies, live birth with minor congenital anomaly(ies), live birth with at least 1 major congenital anomaly, fetal death/still birth with no congenital anomalies, fetal death/still birth with at least 1 major congenital anomaly and unknown outcome (includes participants withdrawn before/at delivery with no available data of pregnancy outcomes).
Time Frame: From Day 1 to Day 42 post-delivery, an average of 2 months
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother
Number analyzed (Participants) | 3557 | 1771
Participants
  Live birth with no congenital anomalies | 3118 | 1555
  Live birth with only minor congenital anomaly(ies) | 317 | 143
  Live birth with at least 1 major congenital anomaly | 61 | 43
  Fetal death/still birth with no congenital anomalies | 9 | 6
  Fetal death/still birth with at least 1 major congenital anomaly | 2 | 0
  Unknown outcome | 50 | 24

36. Secondary Outcome: Number of Maternal Participants With Pregnancy-related Adverse Events of Special Interest (AESIs) From Day 1 to Day 42 Post-delivery
Description: Pregnancy-related AESIs included chorioamnionitis, fetal growth restriction, gestational diabetes mellitus, gestational hypertension, pre-eclampsia, pre-eclampsia with severe features including eclampsia, maternal death, premature preterm rupture of membranes, preterm labor, provider-initiated preterm birth.
Time Frame: From Day 1 to Day 42 post-delivery, an average of 2 months
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother
Number analyzed (Participants) | 3557 | 1771
Participants
  Chorioamnionitis | 30 | 14
  Fetal Growth Restriction | 30 | 26
  Gestational Diabetes Mellitus | 42 | 19
  Gestational Hypertension | 85 | 41
  Pre-Eclampsia | 74 | 36
  Pre-Eclampsia With Severe Features Including Eclampsia | 58 | 28
  Maternal Death | 2 | 1
  Premature Preterm Rupture Of Membranes | 53 | 20
  Preterm Labor | 141 | 57
  Provider-Initiated Preterm Birth | 54 | 16

37. Secondary Outcome: Number of Infant Participants With Neonatal AESIs From Birth to Day 42 Post-birth
Description: Neonatal/infant AESIs included congenital anomalies with functional defects, congenital anomalies with internal structural defects, congenital anomalies with major external structural defects, extremely low birth weight (<1000 grams), low birth weight (<2500 grams), very low birth weight (<1500 grams), neonatal death in a preterm live birth (gestational age >=28 and <37 weeks), neonatal death in a term live birth (>=37 weeks of gestational age), neonatal death in an extremely pre-term birth (gestational age >=22 and <28 weeks), preterm birth (<37 weeks of gestational age), small for gestational age.
Time Frame: From birth to Day 42 post-birth, an average of 2 months
Population: The analysis was performed on the Exposed Set for infants, which included infants live-born to exposed maternal participants, whose parents/LARs completed the informed consent process and signed the informed consent form.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Group - Infant | Placebo Group - Infant
Number analyzed (Participants) | 3494 | 1741
Participants
  Congenital Anomalies With Functional Defects | 5 | 2
  Congenital Anomalies With Internal Structural Defects | 23 | 16
  Congenital Anomalies With Major External Structural Defects | 24 | 14
  Extremely Low Birth Weight (<1000 grams) | 3 | 0
  Low Birth Weight (<2500 grams) | 196 | 102
  Very Low Birth Weight (<1500 grams) | 5 | 0
  Neonatal Death In A Preterm Live Birth (Gestational Age >=28 and <37 Weeks) | 5 | 0
  Neonatal Death In A Term Live Birth (>= 37 Weeks Of Gestational Age) | 6 | 3
  Neonatal Death In An Extremely Pre-Term Birth (Gestational Age >=22 and <28 Weeks) | 2 | 0
  Preterm Birth (<37 Weeks Of Gestational Age) | 237 | 86
  Small For Gestational Age | 253 | 161

ADVERSE EVENTS:
Time Frame: Maternal groups: Solicited AEs - from Day 1 to Day 7 and Unsolicited AEs - from Day 1 to Day 30 post-vaccination. AESIs and MAEs: from Day 1 to Day 42 post-delivery. All-cause mortality, AEs/SAEs leading to withdrawal, SAEs - from Day 1 to Day 181 post-delivery. Infant groups: AESIs: from birth to Day 42 post-birth. All-cause mortality, SAEs, AEs/SAEs leading to withdrawal, MAEs - from birth to Day 366 post-birth.
Description: All events presented in the All-cause mortality, Serious Adverse Events and Other (not including Serious) Adverse Events modules are reported for the Exposed set for maternal participants and Exposed set for infants during the specified time frame.
  The solicited events presented for the RSV MAT Group - Mother and Placebo Group - Mother in the Outcome measures module are reported for the Solicited safety set for maternal participants.
Groups:
- RSV MAT Group - Mother: Maternal participants randomized to the RSV MAT Group received a single dose of the RSV MAT vaccine administered, between 24 to 34 weeks of gestation at Day 1 in this study.
- Placebo Group - Mother: Maternal participants randomized to the Placebo Group received a single dose of placebo administered, between 24 to 34 weeks of gestation, at Day 1 in this study.
Arm/Group | RSV MAT Group - Mother | Placebo Group - Mother | RSV MAT Group - Infant | Placebo Group - Infant
All-Cause Mortality (participants affected / at risk) | 2/3557 | 1/1771 | 20/3494 | 4/1741
Serious Adverse Events (participants affected / at risk) | 827/3557 | 395/1771 | 731/3494 | 371/1741
Other Adverse Events (participants affected / at risk) | 2561/3557 | 1175/1771 | 2615/3494 | 1293/1741
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV MAT Group - Mother (N=3557) | Placebo Group - Mother (N=1771) | RSV MAT Group - Infant (N=3494) | Placebo Group - Infant (N=1741)
ABO incompatibility (Immune system disorders) | 0 (0) | 0 (0) | 7 (7) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 5 (5) | 3 (4) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal labour (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenogenital syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amniorrhoea (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amniotic cavity infection (Infections and infestations) | 12 (12) | 11 (11) | 1 (1) | 0 (0)
Amoebic dysentery (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 11 (11) | 3 (3) | 6 (6) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 9 (9) | 7 (7)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anomalous pulmonary venous connection (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Apgar score low (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aplasia cutis congenita (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Appendicitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 21 (21) | 9 (9) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 22 (22) | 10 (11)
Atrioventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biotinidase deficiency (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood type incompatibility (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Brachycephaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia foetal (Cardiac disorders) | 10 (10) | 4 (4) | 0 (0) | 0 (0)
Bradycardia neonatal (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Brain hypoxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Branchial cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 20 (20) | 5 (5) | 0 (0) | 0 (0)
Brief resolved unexplained event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 56 (61) | 24 (25)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Buried penis syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 8 (8) | 2 (2) | 22 (22) | 10 (11)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) | 1 (1)
Caput succedaneum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carnitine deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 23 (23) | 16 (16) | 0 (0) | 0 (0)
Cerebral cyst (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebral ventricle dilatation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervix dystocia (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 4 (4) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choanal atresia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholestasis of pregnancy (Hepatobiliary disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Chordee (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cleft lip (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cleft lip and palate (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coarctation of the aorta (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congenital cerebral cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Congenital choroid plexus cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Congenital diaphragmatic hernia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital ectopic bladder (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital facial diplegia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital great vessel anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital knee dislocation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital laryngeal stridor (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital melanosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital musculoskeletal disorder of skull (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital myasthenic syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital nephrotic syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital pneumonia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Congenital pyelocaliectasis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital syphilis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Congenital torticollis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Congenital toxoplasmosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniosynostosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Crying (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 16 (16) | 5 (5)
Cyanosis neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystic fibrosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytogenetic abnormality (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death neonatal (General disorders) | 0 (0) | 0 (0) | 13 (13) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 10 (10) | 8 (8)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Developmental delay (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 12 (12) | 9 (10)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dextrocardia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 5 (5)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disseminated neonatal herpes simplex (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmorphism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Dysplasia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ectopic kidney (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometritis (Infections and infestations) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Enlarged clitoris (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epispadias (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythroblastosis foetalis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Exanthema subitum (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face presentation (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Failed forceps delivery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 27 (27) | 12 (12) | 0 (0) | 0 (0)
Failed trial of labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
False labour (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 7 (7) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeding disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibromatosis colli of infancy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foetal anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foetal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal damage (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Foetal disorder (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 125 (125) | 69 (69) | 0 (0) | 0 (0)
Foetal dystocia (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Foetal exposure during delivery (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 17 (17) | 13 (13) | 0 (0) | 0 (0)
Foetal heart rate abnormal (Investigations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Foetal heart rate deceleration abnormality (Cardiac disorders) | 11 (11) | 5 (5) | 0 (0) | 0 (0)
Foetal heart rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 2 (2) | 0 (0) | 0 (0)
Foetal macrosomia (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 3 (3) | 0 (0) | 0 (0)
Foetal malposition (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Foetal monitoring abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fontanelle bulging (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture of clavicle due to birth trauma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fractured skull depressed (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1) | 9 (9) | 7 (7)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital labial adhesions (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genitalia external ambiguous (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 2 (2) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 46 (46) | 22 (22) | 0 (0) | 0 (0)
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Granulosa cell tumour of the testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gynaecological examination abnormal (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Heart disease congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis B surface antigen positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heterotaxia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
High foetal head (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
High risk infant (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hydrops foetalis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 26 (26) | 14 (14)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertelorism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 27 (27) | 9 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypospadias (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 9 (9) | 6 (6)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Hypothermia neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypoxic ischaemic encephalopathy neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Infant irritability (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Infantile colic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infantile haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infantile spasms (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Intestinal malrotation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Iris coloboma (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 89 (91) | 51 (51)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Kernicterus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney duplex (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Labour complication (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leishmaniasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 53 (53) | 21 (21)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macrocephaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Macrosomia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Macrostomia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Male genital examination abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Mastitis (Infections and infestations) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Mastitis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Maternal death (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Measles (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 10 (10) | 8 (8)
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 15 (15) | 6 (6) | 0 (0) | 0 (0)
Medical observation (Investigations) | 1 (1) | 2 (2) | 6 (6) | 3 (3)
Medically induced preterm birth (Surgical and medical procedures) | 37 (37) | 12 (12) | 0 (0) | 0 (0)
Melanoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Menkes' syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metapneumovirus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Microcephaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micrognathia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micropenis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Microtia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Monoplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple congenital abnormalities (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myotonic dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Necrotising colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Neonatal hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Neonatal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Neonatal pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
Neonatal pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 66 (66) | 31 (31)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 23 (23) | 7 (7)
Neonatal seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Newborn persistent pulmonary hypertension (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nonreassuring foetal heart rate pattern (Cardiac disorders) | 19 (19) | 7 (7) | 0 (0) | 0 (0)
Norovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 2 (2) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophageal atresia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 19 (19) | 14 (14) | 0 (0) | 0 (0)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ophthalmia neonatorum (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteochondrodysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteogenesis imperfecta (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papilloma viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 3 (3) | 8 (8)
Pectus excavatum (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 7 (7) | 2 (2)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic haematoma obstetric (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile torsion (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Penoscrotal fusion (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripartum cardiomyopathy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pilonidal disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Placental polyp (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1) | 46 (53) | 21 (22)
Pneumonia adenoviral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 9 (9) | 2 (2)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polydactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (4)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Poor sucking reflex (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 46 (47) | 26 (27) | 0 (0) | 0 (0)
Postpartum sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 105 (106) | 51 (52) | 0 (0) | 0 (0)
Precipitate labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 84 (84) | 30 (30)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 56 (56) | 15 (15) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 5 (5) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 8 (8) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 37 (37) | 14 (14) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 66 (66) | 43 (43) | 0 (0) | 0 (0)
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 7 (7) | 0 (0) | 0 (0)
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 3 (3) | 0 (0) | 0 (0)
Puerperal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Puerperal pyrexia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary venous hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Pyelonephritis (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 3 (3)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 10 (10) | 6 (6)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal disorder in pregnancy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal hypoplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renovascular hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory depth decreased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 19 (19) | 15 (15)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 3 (3) | 0 (0) | 0 (0)
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinoblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinopathy of prematurity (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retrognathia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhesus incompatibility (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Right ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scaphocephaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
Seizure like phenomena (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 46 (46) | 18 (19)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shone complex (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shortened cervix (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Shoulder dystocia (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Skin hypoplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 21 (21) | 15 (15)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 6 (6) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subependymal cyst (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sudden infant death syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supravalvular aortic stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Syndactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syringomyelia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tachycardia foetal (Cardiac disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 7 (7) | 1 (1)
Tethered cord syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thalassaemia alpha (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 28 (30) | 15 (15) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroglossal cyst infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 37 (37) | 16 (16)
Transverse presentation (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Traumatic delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Umbilical cord compression (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Umbilical haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 4 (4)
Urachal abnormality (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urachal sinus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 14 (14) | 11 (11) | 25 (28) | 5 (5)
Urinary tract infection neonatal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine atony (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Uterine cervical laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Uterine hypertonus (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine hypotonus (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 12 (12) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Wound haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wound sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV MAT Group - Mother (N=3557) | Placebo Group - Mother (N=1771) | RSV MAT Group - Infant (N=3494) | Placebo Group - Infant (N=1741)
Anaemia (Blood and lymphatic system disorders) | 62 (62) | 24 (24) | 33 (34) | 12 (12)
Anaemia neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 14 (14) | 5 (5) | 0 (0) | 0 (0)
Bandaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic disease of newborn (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 14 (14) | 5 (5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 6 (6) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Bradycardia foetal (Cardiac disorders) | 7 (7) | 4 (4) | 2 (2) | 0 (0)
Bradycardia neonatal (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Foetal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal heart rate deceleration abnormality (Cardiac disorders) | 7 (7) | 4 (4) | 0 (0) | 1 (1)
Left ventricular dilatation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nonreassuring foetal heart rate pattern (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 6 (6) | 2 (2) | 0 (0) | 1 (1)
Tachycardia foetal (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accessory auricle (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Albinism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 51 (51) | 23 (23)
Anomaly of external ear congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Birth mark (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Carnitine-acylcarnitine translocase deficiency (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cleft uvula (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital hypothyroidism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital melanosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital musculoskeletal disorder of skull (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital naevus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Congenital renal cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 7 (7) | 3 (3)
Congenital syphilis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital thymus absence (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 42 (42) | 21 (21)
Craniosynostosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Cystic fibrosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibromatosis colli of infancy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 11 (11) | 1 (1)
Heart disease congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 11 (11) | 5 (5)
Labial tie (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 6 (6) | 2 (2)
Low set ears (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphatic malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Naevus flammeus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 7 (7) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 7 (7) | 2 (2)
Polydactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Preauricular cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Sickle cell disease (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stahl's ear (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thalassaemia alpha (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 4 (5) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Precocious puberty (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid dysfunction in pregnancy (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transient neonatal hyperthyrotropinaemia (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amblyopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 6 (6) | 2 (2)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 10 (10) | 12 (13)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema eyelids (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 4 (4) | 8 (8)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Orbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trichiasis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 508 (512) | 235 (241) | 22 (22) | 11 (11)
Abdominal pain lower (Gastrointestinal disorders) | 20 (22) | 7 (8) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 3 (3) | 1 (1) | 1 (1)
Allergic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal eczema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal rash (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (12) | 5 (5) | 64 (66) | 23 (24)
Constipation neonatal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 357 (361) | 187 (187) | 97 (107) | 41 (44)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 15 (15) | 5 (6) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enlarged uvula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophilic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 11 (12) | 6 (6)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (9) | 12 (12) | 76 (78) | 46 (48)
Gastrooesophageal reflux in neonate (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gingival cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 21 (22) | 8 (9) | 0 (0) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infantile colic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 15 (15) | 12 (12)
Infantile spitting up (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Meconium plug syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 606 (613) | 307 (313) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic floor dysfunction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 11 (11) | 6 (6)
Tooth demineralisation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth development disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 15 (15) | 8 (8)
Vomiting (Gastrointestinal disorders) | 287 (291) | 153 (153) | 49 (51) | 26 (26)
Vomiting projectile (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Administration site erythema (General disorders) | 133 (136) | 8 (8) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 1294 (1297) | 231 (231) | 0 (0) | 0 (0)
Administration site swelling (General disorders) | 96 (96) | 8 (8) | 0 (0) | 0 (0)
Adverse food reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 6 (7) | 5 (5) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Crying (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Developmental delay (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1094 (1104) | 479 (480) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever neonatal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
High-pitched crying (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypertrophy (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Illness (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (3) | 3 (3) | 9 (14) | 4 (5)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 4 (4) | 1 (1) | 1 (2) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability postvaccinal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macrosomia (General disorders) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 7 (7) | 4 (4) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 43 (44) | 15 (15) | 129 (134) | 53 (60)
Scar inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Swelling face (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholestasis of pregnancy (Hepatobiliary disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 27 (27) | 14 (14)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ABO incompatibility (Immune system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to chemicals (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergy to vaccine (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alloimmunisation (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atopy (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 14 (14) | 6 (6)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0) | 7 (7) | 3 (3)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 18 (18) | 6 (6)
Multiple allergies (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhesus incompatibility (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1) | 2 (2) | 29 (34) | 13 (15)
Acute sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 5 (6) | 4 (4)
Adenoviral upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Amniotic cavity infection (Infections and infestations) | 18 (18) | 3 (3) | 0 (0) | 0 (0)
Amoebic dysentery (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascariasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic bacteriuria (Infections and infestations) | 2 (3) | 4 (4) | 1 (1) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 27 (27) | 7 (7) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 12 (12) | 2 (2) | 0 (0) | 0 (0)
Bacterial vulvovaginitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Balanitis candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bartholin's abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 5 (5) | 5 (5) | 1 (1) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 6 (6)
Breast abscess (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 298 (387) | 152 (175)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 82 (97) | 38 (43)
Bullous impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 117 (118) | 50 (50) | 159 (161) | 90 (90)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 4 (4) | 3 (3) | 16 (17) | 10 (11)
Candida nappy rash (Infections and infestations) | 0 (0) | 0 (0) | 9 (10) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 4 (4) | 0 (0) | 141 (148) | 61 (71)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 11 (11) | 6 (6)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 24 (28) | 12 (13)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dacryocystitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis infected (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dermatophytosis of nail (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Ear infection (Infections and infestations) | 2 (2) | 1 (1) | 120 (148) | 63 (83)
Ear infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema impetiginous (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Endometritis (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema infectiosum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 0 (0) | 0 (0) | 16 (16) | 12 (12)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Eye infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) | 3 (3)
Fungal skin infection (Infections and infestations) | 2 (2) | 0 (0) | 16 (16) | 8 (9)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 13 (13) | 3 (3) | 104 (119) | 60 (68)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 6 (6) | 0 (0) | 14 (15) | 5 (5)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital infection female (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gonococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 38 (38) | 12 (12)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Herpes simplex (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Human herpesvirus 6 infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 27 (27) | 11 (11)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 7 (7) | 3 (3) | 24 (24) | 14 (14)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 45 (51) | 16 (17)
Laryngotracheitis obstructive (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 124 (144) | 60 (72)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 8 (8) | 7 (7)
Mastitis (Infections and infestations) | 42 (42) | 15 (17) | 0 (0) | 0 (0)
Mastitis postpartum (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Metapneumovirus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail bed infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 38 (41) | 19 (20) | 590 (1121) | 306 (557)
Neonatal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neonatal pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Norovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Ophthalmia neonatorum (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 51 (57) | 30 (34)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 2 (2)
Oral viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Otitis externa fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 1 (1) | 114 (141) | 59 (79)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 98 (113) | 45 (55)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Otosalpingitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Parasitic gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Perineal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (5) | 1 (1) | 39 (40) | 14 (14)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 9 (10) | 4 (4)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 31 (31) | 10 (10)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 10 (10) | 3 (3) | 0 (0) | 0 (0)
Puerperal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Puerperal pyrexia (Infections and infestations) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 4 (6) | 3 (3)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 22 (23) | 25 (25)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 34 (34) | 18 (18)
Respiratory tract infection (Infections and infestations) | 51 (55) | 18 (20) | 140 (243) | 65 (131)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 6 (7)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 86 (96) | 46 (50)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 10 (12) | 3 (3)
Roseola (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Scarlet fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 7 (8) | 4 (4) | 9 (9) | 6 (8)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 8 (8)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 2 (4)
Subglottic laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 10 (10) | 4 (4) | 59 (61) | 18 (19)
Syphilis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Systemic viral infection (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 2 (3)
Thyroglossal cyst infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea capitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1) | 14 (14) | 8 (8)
Tooth abscess (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxoplasmosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 71 (86) | 37 (43) | 848 (1703) | 396 (779)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 104 (107) | 49 (50) | 29 (32) | 9 (9)
Urogenital infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vaccination site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 9 (9) | 3 (3) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 8 (8) | 4 (4)
Viral diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 36 (37) | 12 (12)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 22 (22) | 11 (11)
Viral rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 43 (55) | 24 (37)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 13 (13) | 9 (9) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 6 (6) | 5 (5) | 0 (0) | 0 (0)
Vulvovaginitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginitis trichomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Wound sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental exposure to product packaging (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Anal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4) | 3 (4)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone fissure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chemical burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 5 (5) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 7 (7) | 5 (5)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body ingestion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture of clavicle due to birth trauma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 9 (9) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Incision site dermatitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site rash (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Perineal injury (Injury, poisoning and procedural complications) | 71 (71) | 37 (37) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post vaccination fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Radial head dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 3 (3) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral injury (Injury, poisoning and procedural complications) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Uterine cervical laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 45 (45) | 18 (18) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acoustic stimulation tests abnormal (Investigations) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Apgar score low (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Audiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Blood glucose increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Blood iron decreased (Investigations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 5 (5) | 6 (6) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 28 (28) | 11 (11)
Cardiac murmur functional (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coombs direct test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coombs test positive (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Drug screen positive (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Electroencephalogram normal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foetal heart rate abnormal (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Foetal heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal heart rate indeterminate (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Foetal monitoring (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal monitoring abnormal (Investigations) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Foetal non-stress test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HIV test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Head circumference abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Human rhinovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immunoreactive trypsinogen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza A virus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inhibin A increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kleihauer-Betke test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical observation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otoacoustic emissions test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin B12 decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast milk substitute intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (6)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dairy intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 17 (17) | 10 (10)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 9 (9) | 4 (4) | 1 (1) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Milk soy protein intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Overweight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
Poor feeding infant (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 12 (13) | 3 (4)
Underweight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 6 (6)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (7) | 2 (2)
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 21 (21) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Asymmetric gluteal fold (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Asymmetric thigh fold (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (22) | 11 (11) | 0 (0) | 0 (0)
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone hypertrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Head deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Hypertonia neonatal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotonia neonatal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint laxity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint noise (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament laxity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Newborn head moulding (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nose deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pubic pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Short stature (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Snapping hip syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 10 (10) | 2 (2)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infantile haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ulcerated haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Xanthogranuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Fontanelle depressed (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gross motor delay (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 962 (993) | 452 (465) | 0 (0) | 0 (0)
Hypertonia (Nervous system disorders) | 0 (0) | 0 (0) | 8 (8) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 8 (9) | 4 (4)
IVth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infant irritability (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Language disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Motor developmental delay (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Movement disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurodevelopmental delay (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Seizure like phenomena (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subependymal cyst (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tethered cord syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal cord insertion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Afterbirth pain (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amniorrhexis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amniorrhoea (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Birth trauma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 9 (10) | 3 (3) | 0 (0) | 0 (0)
Caput succedaneum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 7 (7) | 3 (3)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 10 (10) | 4 (4)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Complication of delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 6 (6) | 0 (0) | 0 (0)
Face presentation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
False labour (Pregnancy, puerperium and perinatal conditions) | 5 (6) | 4 (4) | 0 (0) | 0 (0)
Foetal acidosis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foetal damage (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 18 (18) | 6 (7) | 0 (0) | 0 (0)
Foetal dystocia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 16 (16) | 15 (15) | 0 (0) | 0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 18 (19) | 7 (7) | 0 (0) | 0 (0)
Foetal macrosomia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 35 (35) | 18 (18) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 42 (42) | 20 (20) | 0 (0) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothermia neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intrapartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 207 (207) | 70 (70)
Labour complication (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Labour pain (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 9 (9) | 9 (9)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 151 (151) | 82 (82)
Meconium abnormal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 5 (5) | 3 (3) | 0 (0)
Meconium stain (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Neonatal disorder (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 25 (25) | 10 (10) | 0 (0) | 0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Placental calcification (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Placental disorder (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Placental polyp (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 7 (8) | 4 (4) | 0 (0) | 0 (0)
Poor weight gain neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 32 (32) | 22 (22) | 0 (0) | 0 (0)
Postpartum uterine subinvolution (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 25 (25) | 11 (11) | 0 (0) | 0 (0)
Precipitate labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 153 (153) | 56 (56)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 84 (84) | 43 (43) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 4 (4) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 17 (17) | 6 (6) | 0 (0) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 6 (6) | 0 (0) | 0 (0)
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 3 (3) | 0 (0) | 0 (0)
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shoulder dystocia (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 3 (3) | 4 (4) | 2 (2)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 233 (233) | 147 (147)
Subchorionic haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Transverse presentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 0 (0) | 3 (3) | 1 (1)
Umbilical cord compression (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical cord haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 12 (12) | 4 (4)
Uterine atony (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 10 (11) | 0 (0) | 0 (0)
Uterine hypertonus (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine hypotonus (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Uterine inversion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine irritability (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 7 (7) | 3 (3) | 0 (0) | 0 (0)
Brief psychotic disorder, with postpartum onset (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perinatal depression (Psychiatric disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Postpartum anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychomotor retardation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Selective eating disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Tearfulness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atonic urinary bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Vesicoureteric reflux (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bilateral breast buds (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast engorgement (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Breast inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coital bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital blister (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital labial adhesions (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 8 (8) | 3 (3)
Genital macule (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital ulceration (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Lactation disorder (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Lactation insufficiency (Reproductive system and breast disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Nipple disorder (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Penile adhesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shortened cervix (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular retraction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Threatened uterine rupture (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine scar (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 14 (15) | 7 (8) | 1 (1) | 2 (2)
Vaginal disorder (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 17 (17) | 1 (1) | 1 (1) | 0 (0)
Vulval oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 8 (8) | 6 (6)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brief resolved unexplained event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 8 (9) | 4 (4)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 20 (31) | 5 (6)
Bronchiolitis obliterans syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 12 (14) | 10 (12)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 7 (11) | 6 (9)
Childhood asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (4) | 180 (251) | 82 (109)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 18 (21) | 13 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immature respiratory system (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 142 (160) | 57 (64)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (7) | 4 (4)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (8) | 2 (2)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neonatal respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 12 (12) | 7 (7)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 0 (0) | 2 (2)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (5) | 1 (1)
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5) | 141 (343) | 72 (162)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 19 (21) | 7 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 120 (191) | 51 (80)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 12 (12) | 8 (8)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 7 (8) | 7 (11)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 23 (24) | 15 (16)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 7 (7) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cellulite (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 35 (35) | 15 (15)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 56 (58) | 42 (44)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 10 (10) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 113 (124) | 55 (58)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 76 (76) | 34 (37)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (4)
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes gestationis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Melanoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 33 (35) | 15 (15)
Nail fold inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pityriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polymorphic eruption of pregnancy (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prurigo of pregnancy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 5 (5) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 53 (53) | 24 (27)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Rash neonatal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 72 (72) | 27 (27)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Transient neonatal pustular melanosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Umbilical discharge (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 6 (6) | 2 (2)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Episiotomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medically induced preterm birth (Surgical and medical procedures) | 17 (17) | 4 (4) | 0 (0) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyanosis (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 13 (13) | 11 (11) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 7 (7) | 3 (3) | 0 (0) | 1 (1)
Inferior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vasodilatation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT04605159/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT04605159/SAP_001.pdf